CLINICAL TRIAL: NCT00714272
Title: Therapeutic Effect of Granulocytapheresis in Psoriasis (GRIP-study)Using a Novel Cellulose-based Adsorber Device
Brief Title: Granulocytapheresis in Psoriasis
Acronym: GRIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary outcome not achieved.
Sponsor: EXcorLab GmbH (Other)
Collaborators: Membrana GmbH (Industry); Nikkiso Co. Ltd (Industry); Nikkiso Medical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KSGA0801; F002MN0107_1
Record Dates: First submitted 2008-06-04; First posted 2008-07-14 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-07

CONDITIONS: Psoriasis
Keywords: granulocytapheresis, psoriasis, PASI, apheresis
MeSH Terms: conditions — Psoriasis | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Granulocytapheresis treatment
  Interventions: Device: Treatment with a Granulocyte Adsorber, Medica Adsorber 1.1
- B (Placebo Comparator): Sham device treatment
  Interventions: Device: Treatment with a sham device, EXcorLab box 1.2

INTERVENTIONS:
Device: Treatment with a Granulocyte Adsorber, Medica Adsorber 1.1 — 6 treatments. One per week during the first six consecutive weeks.
  Arms: A
Device: Treatment with a sham device, EXcorLab box 1.2 — 6 sham treatments. One treatment per week during the first six consecutive weeks.
  Arms: B

SUMMARY:
In a prospective, randomized, controlled, double-blinded, multicenter study, granulocytapheresis using a novel cellulose-based adsorber will be compared to control sham treatment (placebo). The effects on clinical symptoms and on some inflammatory parameters of patients with moderate to severe plaque psoriasis will be evaluated over a 24-week period.

The primary end-point is a ≥75 percent improvement in PASI (Psoriasis Area and Severity Index).

The study purpose is to demonstrate a beneficial therapeutic effect of granulocytapheresis using the novel cellulose-based adsorber device in moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe plaque psoriasis with a PASI >/=10
* Age >/= 18 years
* Negative pregnancy test in woman of childbearing age acceptable method of contraception for both men and women
* Written informed consent that can be withdrawn at any time or for any reason
* Discontinuation of any systemic psoriasis treatment. Washout period of at least two weeks for prior systemic medications
* Only emollients for topical treatment
* No vaccinations for at least 14 days prior to first treatment

Exclusion Criteria:

* Other forms of psoriasis (e.g., guttate, pustular, erythrodermic, palmoplantar etc.)
* History of ongoing uncontrolled bacterial, fungal or viral infection (including opportunistic infections); HIV positivity
* Pregnancy
* Clinically relevant thrombocytopenia or bleeding disorders
* WBC <4.000 or >12.000/µl
* Malignancy within the last five years (exception: successfully treated basal cell carcinoma or squamous cell carcinoma of the skin)
* Severe cardiac disorders, stroke, pulmonary disease within the last year
* Any medical condition that, in the judgment of the investigators, would jeopardize the patient's safety during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-02-18 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Schoen, Prof.Dr.med., Principal Investigator — University of Goettingen, Department of Dermatology and Venerology; Christoph Wanner, Prof.Dr.med., Study Director — University Hospital Wuerzburg, Department of Medicine; Eva B Broecker, Prof.Dr.med., Study Director — University of Wuerzburg, Department of Dermatology; Gerhard A Mueller, Prof.Dr.med., Study Director — University of Goettingen, Department of Nephrology and Rheumatology; Detlef Krieter, Dr.med., Study Director — University Hospital Wuerzburg, Department of Medicine
Locations (2):
- Germany (2):
  - University of Würzburg, Department of Medicine, Division of Nephrology, and Department of Dermatology, Würzburg, Bavaria
  - University of Göttingen, Department of Dermatology and Department of Nephrology and Rheumatology, Göttingen, Lower Saxony

RESULTS

PARTICIPANT FLOW:
Groups:
- A - Verum, Granulocytapheresis: Granulocytapheresis treatment
  Treatment with a Granulocyte Adsorber, Medica Adsorber 1.1: 6 treatments. One per week during the first six consecutive weeks.
- B - Control, Sham Treatment: Sham device treatment
  Treatment with a sham device, EXcorLab box 1.2: 6 sham treatments. One treatment per week during the first six consecutive weeks.
Period: Overall Study
Arm/Group | A - Verum, Granulocytapheresis | B - Control, Sham Treatment
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A - Verum, Granulocytapheresis | B - Control, Sham Treatment | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 40.5 [28 to 63] | 49.5 [43 to 56] | 45 [28 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: >/=75 % Improvement in PASI (Psoriasis Area and Severity Index) on an Intention-to-treat Basis
Time Frame: At the end of the granulocytapheresis treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | A - Verum, Granulocytapheresis | B - Control, Sham Treatment
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

2. Secondary Outcome: Patients Achieving an Improvement of PASI by >/= 50%
Time Frame: From baseline to weeks 2, 6, 12 and 24
Measure: Count of Participants; unit: Participants
Arm/Group | A - Verum, Granulocytapheresis | B - Control, Sham Treatment
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | A - Verum, Granulocytapheresis | B - Control, Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - Verum, Granulocytapheresis (N=2) | B - Control, Sham Treatment (N=2)
Nausea (General disorders) | 1 (2) | 1 (3)

LIMITATIONS AND CAVEATS:
The study was discontinued after only 4 patients because of unforeseen exit of PI from the study location.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No